CLINICAL TRIAL: NCT03648996
Title: Sex-related Differences in Arterial Stiffness in Type 2 Diabetics: Role of Uric Acid
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Camila Manrique, MD, Associate Professor of Medicine, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012106
Record Dates: First submitted 2018-08-16; First posted 2018-08-28 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus, Type 2; Hyperuricemia
Keywords: arterial stiffness; endothelial dysfunction; type 2 diabetes; hyperuricemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperuricemia | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Low-fructose diet, isocaloric (Experimental): Subjects assigned to this arm of the study will consume for 6 months a diet low in fructose while maintaining baseline body weight.
  Interventions: Other: Low-fructose diet, isocaloric
- Allopurinol (Experimental): Subjects assigned to this arm of the study will be treated for 6 months with allopurinol (max dose 300 mg)
  Interventions: Drug: Allopurinol
- Placebo (Placebo Comparator): Subjects assigned to this arm will receive placebo
  Interventions: Drug: Placebo
- Low-fructose diet, hypocaloric (Experimental): Subjects assigned to this arm of the study will consume for 6 months a diet low in fructose with a 500 Calorie energy reduction.
  Interventions: Other: Low-fructose, hypocaloric

INTERVENTIONS:
Other: Low-fructose diet, isocaloric — 6 month of consumption a low fructose diet
  Arms: Low-fructose diet, isocaloric
Drug: Allopurinol — 6 months of allopurinol treatment with the goal of decreasing uric acid compared to control group
  Other Names: Zyloprim
  Arms: Allopurinol
Drug: Placebo — 6 months of placebo treatment
  Arms: Placebo
Other: Low-fructose, hypocaloric — 6 month of consumption a low fructose diet with a 500 Calorie/day energy restriction
  Arms: Low-fructose diet, hypocaloric

SUMMARY:
Three separate interventions will be undertaken with the primary outcome of improving pulse wave velocity. Initially, age and BMI-matched men and post-menopausal women, all with type 2 diabetes, will be treated with allopurinol (20 men, 20 women) for 6 months, in order to reduce serum uric acid (SUA) concentrations relative to placebo (10 men, 10 women). In a second intervention, dietary fructose will be restricted for a period of 6 months in type 2 diabetes (T2D) subjects who will maintain a stable weight (20 men, 20 women). In a third intervention, dietary fructose will be restricted for a period of 6 months in type 2 diabetes (T2D) subjects who will achieve a caloric deficit and weight reduction (20 men, 20 women). At the beginning and end of each of the studies, measures of arterial stiffness will be combined with assessments of endothelial function (flow-mediated dilation and insulin stimulated leg blood flow), measurements of systemic inflammation and oxidative stress.

DETAILED DESCRIPTION:
Sedentary, overweight and obese subjects diagnosed with T2D, ages 40-75 years old, will be recruited from the local community, via the University of Missouri's Endocrinology Clinic and the primary care clinics. During screening, and after consent, anthropometrics (waist circumference and body composition) will be obtained and fasting blood will be drawn for serum chemistries, A1c, complete blood count, liver and kidney function. Screening will also include completion of an oral glucose tolerance test with measurements of arterial stiffness and assessment of endothelial function. Following screening, eligible subjects will be assigned to one of the four groups (allopurinol, placebo, fructose restriction/isocaloric, or fructose restriction/hypocaloric). Allopurinol will be titrated to achieve a target dose of 300 mg/day. Along with placebo, this arm of the study is double-blinded. A separate group of men and women will be assigned to the isocaloric fructose-restriction study in which dietary fructose is replaced by starch and body weight is held constant. Lastly, a separate group of men and women will be assigned to the hypocaloric fructose-restriction in which baseline caloric intake will be reduced by 500 Calories/day while baseline intakes of protein and fat will remain constant. The subjects in these groups will not be blinded to the dietary treatment but the staff making measurements will be. Subjects in the four groups will be matched for age and BMI.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 40-75 years at randomization
* BMI between 25.1 and 50 kg/m2.
* Type 2 diabetes diagnosed > 3 months ago. Patients with T2D will be classified based on physician diagnosis.

Exclusion Criteria:

* serum uric acid < 5.5 mg/dL (for medication/allopurinol and isocaloric low-fructose diet arm)
* habitual diet containing low amount of sugars < 5% of total energy intake
* recent CVD event (stroke, heart failure hospitalization, revascularization or acute coronary event in the last 12 months).
* abnormal thyroid tests or chronic liver disease
* stage IV renal disease (GFR <30)
* hyperparathyroidism
* use of azathioprine
* active cancer
* autoimmune diseases
* excessive alcohol consumption (>14 drinks/week for men, >7 drinks/week for women)
* current tobacco use
* bodyweight change ≥10% within the last 6 months
* history of gout or uncontrolled hypertension
* A1C >10 % (only for medication/placebo arm)
* Pregnancy or lactation in women (or women not using contraceptives)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Camila Manrique Acevedo, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The current Clinical trials.gov information reflects the number of subjects that were recruited for the clinical trial portion of this study. No subjects were recruited the isocaloric portion of this study.
Period: Overall Study
Arm/Group | Allopurinol | Placebo | Low-fructose Diet, Hypocaloric
Started | 9 | 7 | 18
Completed | 7 | 5 | 16
Not Completed | 2 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 2
Not completed — Physician Decision | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Allopurinol | Placebo | Low-fructose Diet, Hypocaloric | Total
Number analyzed (Participants) | 7 | 5 | 16 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9 | 18
  >=65 years | 2 | 1 | 7 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (8.6) | 58 (7.5) | 59 (12.1) | 59 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 9 | 15
  Male | 4 | 2 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 5 | 15 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 5 | 16 | 28
Baseline PWV [Mean (Standard Deviation); unit: m/s] — Assessment of arterial stiffness, carotid femoral pulse wave velocity Population: Measurement not available in all participants
  m/s
    number analyzed (Participants) | 7 | 5 | 15 | 27
    (all) | 9.87 (3.36) | 8.62 (1.45) | 8.17 (1.19) | 8.7 (2.06)
Brachial FMD [Mean (Standard Deviation); unit: Percentage (%)] — Population: Measurement not available in all participants
  Percentage (%)
    number analyzed (Participants) | 7 | 5 | 13 | 25
    (all) | 4.75 (3.37) | 4.29 (0.77) | 5.15 (3.14) | 4.86 (2.83)

OUTCOME MEASURES:

1. Primary Outcome: Carotid Femoral Pulse Wave Velocity (cfPWV)
Description: It is the gold standard non-invasive index of arterial stiffness. Transit time between carotid and femoral pressure waves is calculated using the foot-to-foot method. cfPWV is calculated as distance traveled by the pulse wave (i.e., femoral location-sternal notch minus sternal notch-carotid location) divided by pulse transit time. All the measurements will be done by the same blinded technician
Time Frame: This will be assessed at baseline and 6 months (final). The goal is to assess changes from baseline when compared to final time point.
Population: Measurement not available for all subjects
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Allopurinol | Placebo | Low-fructose Diet, Hypocaloric
Number analyzed (Participants) | 6 | 4 | 15
m/s | 8.71 (1.47) | 7.8 (1.04) | 8.28 (1.40)

2. Secondary Outcome: Brachial Artery Flow Mediated Dilation (FMD)
Description: Brachial artery FMD will be assessed at baseline and final. FMD is a measurement of conduit artery endothelial function. FMD is assessed immediately after each PWV measurement. Shear rate AUC until peak diameter is calculated as stimulus for FMD and used in covariate analysis as described. All measurements will be performed, under co-I supervision by the same blinded technician.
Time Frame: Baseline and 6 months (final). The goal is to assess changes from baseline when compared to final time point.
Population: Measurement not available for all subjects
Measure: Mean (Standard Deviation); unit: Percentage (%)
Groups:
- Allopurinol: Allopurinol 6 mo
- Placebo: Placebo 6-mo
- Low-fructose Diet, Hypocaloric: Low-fructose diet, hypocaloric 6 mo
Arm/Group | Allopurinol | Placebo | Low-fructose Diet, Hypocaloric
Number analyzed (Participants) | 7 | 5 | 16
Percentage (%) | 5.03 (3.44) | 4.4 (2.8) | 7.10 (2.19)

3. Secondary Outcome: Insulin-stimulated Leg Blood Flow
Description: We will perform a hyperinsulinemic euglycemic clamp to evaluate insulin-stimulated leg blood flow (to be assessed via Doppler ultrasound). Insulin will be infused at a constant rate to mimic postprandial insulin concentrations and glucose maintained at fasting values via a variable 20% dextrose infusion. Femoral artery blood flow will be assessed at the beginning and at end of the 60-minute insulin infusion, and data are presented as percent of change from pre-insulin infusion values.
Time Frame: The goal is to assess insulin stimulated responses in blood flow after 6 mo of intervention.
Population: The percentage change in blood flow in response to insulin was calculated as femoral blood flow insulin - femoral blood flow insulin no insulin x 100
Measure: Mean (Standard Deviation); unit: Percetage (%) change
Arm/Group | Allopurinol | Placebo | Low-fructose Diet, Hypocaloric
Number analyzed (Participants) | 7 | 5 | 11
Percetage (%) change | -7.68 (35.29) | 68.18 (153.59) | 42.65 (75.12)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Subjects enrolled in the allopurinol/placebo arm were administered a safety formulary at weeks 2, 4, 6, 8,12, 16, and 20 to assess for common side effects.
  Subjects in the hypocaloric arm were contacted by the research team weekly from week 1 thru 6, and then at week 8, 12, 16, and 20 to assess for any changes in their health
Arm/Group | Allopurinol | Placebo | Low-fructose Diet, Hypocaloric
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5 | 1/16
Other Adverse Events (participants affected / at risk) | 5/7 | 4/5 | 8/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allopurinol (N=7) | Placebo (N=5) | Low-fructose Diet, Hypocaloric (N=16)
Urinary tract infection/pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — hospital admission
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Allopurinol (N=7) | Placebo (N=5) | Low-fructose Diet, Hypocaloric (N=16)
Diarrhea (Gastrointestinal disorders) | 4 | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 0
Skin rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Non severe hypoglycemia (Endocrine disorders) | 0 | 0 | 5
Glucosuria (Endocrine disorders) | 0 | 0 | 1
Ankle Sprain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Acid Reflux (Gastrointestinal disorders) | 0 | 0 | 1
Severe hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The covid pandemic limited recruitment efforts. Protocol was modified to limit the risk of exposure of research staff and research participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/96/NCT03648996/Prot_SAP_000.pdf
  • Informed Consent Form: General (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/96/NCT03648996/ICF_001.pdf
  • Informed Consent Form: Allopurinol/Placebo Arm (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/96/NCT03648996/ICF_002.pdf
  • Informed Consent Form: Hypocaloric Low Fructose Diet Arm (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/96/NCT03648996/ICF_003.pdf